CLINICAL TRIAL: NCT04727008
Title: Phase I Study of A CXCR4 Modified BCMA CAR-T in Patients With Refractory and/or Relapsed Multiple Myeloma
Brief Title: CXCR4 Modified Anti-BCMA CAR T Cells for Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Ting Niu, Director of Department of Hematology, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCART-001
Record Dates: First submitted 2020-11-30; First posted 2021-01-27 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXCR4 modified anti-BCMA CAR T cell therapy (Experimental): CAR T cell therapy
  Interventions: Biological: CXCR4 modified anti-BCMA CAR T cells

INTERVENTIONS:
Biological: CXCR4 modified anti-BCMA CAR T cells — intravenous infusion

SUMMARY:
Multiple myeloma (MM) is an incurable plasma cell cancer that almost all patients eventually relapse despite advancement in treatment strategies. B-cell maturation antigen (BCMA) is a cell surface receptor that expressed primarily by malignant and normal plasma cells. This study aims to evaluate the safety and tolerance CXCR4 modified BCMA CAR T cells in treating standard treatment failed refractory/relapsed multiple myeloma, and will follow dose-escalating cohorts. The efficacy of CXCR4 modified BCMA CAR T will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 75 years old.
2. The expected survival ≥ 12 week
3. ECOG ≤ 2
4. Patients with multiple myeloma that never achieved MR (minor response) or received ≥ 1 line of standard therapy but tumor relapse
5. The liver and renal function is good/adequate organ function; no uncontrolled or active infectious disease
6. Venous channel is unobstructed, which can meet the needs of intravenous drip; no contraindications of mononuclear cell collection
7. Patients can take effective contraceptive measures during the trial period and 1 year after the infusion
8. Voluntary informed consent is given, agree to follow the trial treatment and visit plan

Exclusion Criteria:

1. Patients with other uncontrollable cancer
2. Active hepatitis B, hepatitis C, or HIV infection
3. Other uncontrolled active disease
4. Patients with coronary heart disease, angina pectoris, myocardial infarction, cerebral thrombosis, cerebral hemorrhage or any other severe diseases
5. Patients with uncontrollable hypertension(≥ grade II)
6. Patients with history of uncontrollable mental illness
7. Long-term use of immunosuppressants after organ transplantation (inhaled corticosteroids are excluded)
8. Unstable pulmonary embolism or any arteriovenous embolism 30 days before enrollment;
9. Pregnant or lactating women; Men or women who have a pregnancy plan within a year; The patients cannot guarantee effective contraceptive measures during the trial period;
10. Patients with uncontrollable infectious disease or need systematic treatment within the 14 days of enrollment;
11. Patients had other conditions that were not appropriate for the study determined by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | 2 years
  Dose Limiting Toxicities (DLTs) during the first 28 days after anti-BCMA CAR-T cell administration
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 24 months

SECONDARY OUTCOMES:
ORR (overall response rate) | 3 months，6 months
  Proportion of subjects with the best overall response (BOR)
CRR (complete response rate) | 3 months
  Proportion of subjects with the BOR of sCR+CR at Month 3

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No